CLINICAL TRIAL: NCT07352501
Title: RCT of Pulsed Electromagnetic Fields Plus Nutraceutical Supplementation in Women With Distal Radius Fracture
Brief Title: Effectiveness of Pulsed Electromagnetic Fields and Nutraceutical Supplementation in Women With Distal Radius Fracture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFR052025
Record Dates: First submitted 2025-12-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Fracture of Distal Radius; Bone Fractures; Wrist Injuries
Keywords: distal radius fracture; wrist injury; pulsed electromagnetic fields; nutraceutical supplementation; bone healing; pain management; functional recovery
MeSH Terms: conditions — Fractures, Bone; Wrist Injuries; Wrist Fractures; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF therapy alone (standard care) (Active Comparator)
  Interventions: Device: Pulsed Electromagnetic Field Therapy
- PEMF therapy + daily nutraceutical supplementation (Experimental)
  Interventions: Device: Pulsed Electromagnetic Field Therapy; Dietary Supplement: Nutraceutical Supplement

INTERVENTIONS:
Device: Pulsed Electromagnetic Field Therapy — 9 hours per day for 30 consecutive days using a wearable PEMF device
Dietary Supplement: Nutraceutical Supplement — Daily oral dose containing vitamin D, vitamin K, magnesium, vitamin C, zinc, and copper for 30 days
  Arms: PEMF therapy + daily nutraceutical supplementation

SUMMARY:
This single-center randomized controlled trial tests whether adding a daily nutraceutical supplement to standard pulsed electromagnetic field (PEMF) therapy improves recovery after a recent distal radius (wrist) fracture in women. The study asks: does PEMF plus a supplement of vitamin D, vitamin K, magnesium, vitamin C, zinc, and copper produce faster bone healing, greater pain relief, less soft-tissue swelling, and fewer complications (including complex regional pain syndrome) than PEMF alone? Sixty women aged 45-55 with a recent radiographically confirmed distal radius fracture and baseline pain NRS ≥ 4 are randomized 1:1. One group receives PEMF 9 hours per day for 30 days. The other group receives the same PEMF regimen plus the daily oral nutraceutical for 30 days. Assessments occur at baseline, 15 days (early ultrasound and laboratory markers), and 30 days (radiographic healing, Budapest criteria for complex regional pain syndrome, pain NRS, and functional measures).

The primary outcomes are change in pain (NRS) and early callus formation at 15 days, with radiographic healing at 30 days. Secondary outcomes include biochemical markers of bone turnover, 24-hour calciuria and phosphaturia, soft-tissue edema by ultrasound, functional recovery, safety, and tolerability. The hypothesis is that the combined treatment leads to earlier and clinically meaningful improvements in pain, function, and bone repair compared with PEMF alone.

DETAILED DESCRIPTION:
This trial investigates whether adding a defined daily nutraceutical regimen to an established pulsed electromagnetic field (PEMF) protocol influences early biological fracture repair and short-term clinical recovery in peri-menopausal women with recent distal radius fractures; it is designed to link biochemical markers, imaging signals, device usage data, and patient-reported outcomes to test the hypothesis that targeted micronutrient support potentiates PEMF-mediated osteogenic and anti-inflammatory effects, accelerating early callus formation, reducing pain and soft-tissue swelling, and maintaining acceptable safety and tolerability. The trial employs centralized randomization, standardized visit windows, and pre-specified procedures for specimen handling, imaging acquisition, and blinded read workflows to ensure temporal comparability and measurement quality; adherence is monitored through device logs, pill counts, and participant diaries, with defined follow-up for nonadherence. Data are captured in source documents and an electronic database with validation checks, role-based access, audit trails, and QA processes including internal monitoring and independent adjudication of discordant imaging reads. The statistical framework follows intention-to-treat principles with mixed-effects models for repeated measures, pre-specified sensitivity and per-protocol analyses, and strategies for handling missing data and potential confounders; subgroup analyses explore baseline nutritional status and device usage intensity. Safety oversight includes continuous adverse event capture, graded severity and causality assessment, and predefined reporting pathways to study safety officers and the ethics committee. Ethical and regulatory compliance adheres to Good Clinical Practice and local regulations, with informed consent, participant confidentiality safeguards, GMP-compliant product handling, and procedures for protocol deviations and safety signals. Results will be reported with effect estimates and confidence intervals, interpreted for clinical relevance and biological coherence across biomarkers and imaging, and disseminated through peer-reviewed publications and lay summaries for participants and stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged
* Radiographically confirmed distal radius fracture within 5 days of trauma
* Presentation to the hospital within 3 days of the fracture event
* Fracture treated conservatively with a cast (non-surgical management)
* Baseline pain score ≥ 4 on the Numeric Rating Scale (NRS)
* Ability to provide informed consent
* Willingness to comply with study procedures and follow-up visits

Exclusion Criteria:

* Bilateral wrist fractures
* Prior surgery on the affected wrist
* Use of bone-active medications (e.g., bisphosphonates, corticosteroids) in the past 6 months
* Known allergy or intolerance to any component of the nutraceutical supplement
* Presence of implanted electronic devices (e.g., pacemaker)
* Cognitive impairment or psychiatric condition interfering with consent or adherence
* Pregnancy or breastfeeding
* Participation in another clinical trial within the past 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Radiographic fracture healing (proportion with cortical bridging) at 30 days | 30 days post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. Paolo Giaccone, Palermo, Italy, Italy